CLINICAL TRIAL: NCT03334422
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Baricitinib in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Study of Baricitinib (LY3009104) in Patients With Moderate to Severe Atopic Dermatitis
Acronym: BREEZE-AD2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16581; I4V-MC-JAHM (Other: Eli Lilly and Company); 2017-000871-10 (EudraCT Number)
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Atopic Dermatitis
Keywords: eczema; atopic eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 4 Milligram (mg) Baricitinib (Experimental): 4mg Baricitinib administered orally once daily. Placebo 1 mg and 2 mg administered orally every day to match
  Interventions: Drug: Baricitinib; Drug: Placebo
- 2mg Baricitinib (Experimental): 2mg Baricitinib administered orally once daily. Placebo 1 mg and 4 mg administered orally every day to match.
  Interventions: Drug: Baricitinib; Drug: Placebo
- 1mg Baricitinib (Experimental): 1mg Baricitinib administered orally once daily. Placebo 2 mg and 4 mg administered orally every day to match.
  Interventions: Drug: Baricitinib; Drug: Placebo
- Placebo (Placebo Comparator): Placebo administered orally once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
  Arms: 1mg Baricitinib; 2mg Baricitinib; 4 Milligram (mg) Baricitinib
Drug: Placebo — Administered orally

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of baricitinib as monotherapy in participants with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with moderate to severe Atopic Dermatitis for at least 12 months.
* Have had inadequate response or intolerance to existing topical (applied to the skin) medications within 6 months preceding screening.
* Are willing to discontinue certain treatments for eczema (such as systemic and topical treatments during a washout period).
* Agree to use emollients daily.

Exclusion Criteria:

* Are currently experiencing or have a history of other concomitant skin conditions (e.g., psoriasis or lupus erythematosus), or a history of erythrodermic, refractory, or unstable skin disease that requires frequent hospitalizations and/or intravenous treatment for skin infections.
* A history of eczema herpeticum within 12 months, and/or a history of 2 or more episode of eczema herpeticum in the past.
* Participants who are currently experiencing a skin infection that requires treatment, or is currently being treated, with topical or systemic antibiotics.
* Have any serious illness that is anticipated to require the use of systemic corticosteroids or otherwise interfere with study participation or require active frequent monitoring (e.g., unstable chronic asthma).
* Have been treated with the following therapies:

  * Monoclonal antibody for less than 5 half-lives prior to randomization.
  * Received prior treatment with any oral Janus kinase (JAK) inhibitor.
  * Received any parenteral corticosteroids administered by intramuscular or intravenous (IV) injection within 2 weeks prior to study entry or within 6 weeks prior to planned randomization or are anticipated to require parenteral injection of corticosteroids during the study.
  * Have had an intra-articular corticosteroid injection within 2 weeks prior to study entry or within 6 weeks prior to planned randomization.
* Have high blood pressure characterized by a repeated systolic blood pressure >160 millimeters of mercury (mm Hg) or diastolic blood pressure >100 mm Hg.
* Have had major surgery within the past eight weeks or are planning major surgery during the study.
* Have experienced any of the following within 12 weeks of screening: venous thromboembolic event (VTE), myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage III/IV heart failure.
* Have a history of recurrent (≥ 2) VTE or are considered at high risk of VTE as deemed by the investigator.
* Have a history or presence of cardiovascular, respiratory, hepatic, chronic liver disease gastrointestinal, endocrine, hematological, neurological, lymphoproliferative disease or neuropsychiatric disorders or any other serious and/or unstable illness.
* Have a current or recent clinically serious viral, bacterial, fungal, or parasitic infection including herpes zoster, tuberculosis.
* Have specific laboratory abnormalities.
* Have received certain treatments that are contraindicated.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (80):
- Argentina (8):
  - CENIT Centro de Neurociencias, Investigación y Tratamiento, Caba, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Clinica Adventista de Belgrano, Ciudad de Buenos Aires, Buenos Aires
  - Fundacion CIDEA, Buenos Aires
  - Instituto de Neumonología y Dermatología, Buenos Aires
  - Psoriahue Medicina Interdisciplinaria, Buenos Aires
  - Buenos Aires Skin, Ciudad Autonoma Buenos Aires
  - Parra Dermatología, Mendoza
- Australia (6):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - Skin & Cancer Foundation Australia, Westmead, New South Wales
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Clinical Trials SA Pty Ltd, Adelaide, South Australia
  - Skin and Cancer Foundation Inc., Carlton, Victoria
  - Fremantle Dermatology, Perth, Western Australia
- Austria (5):
  - Ordensklinikum Linz GmbH - Elisabethinen, Linz, Upper Austria
  - KA Rudolfstiftung, Vienna
  - AKH, Vienna
  - KH Hietzing mit neurologischem Zentrum Rosenhügel, Vienna
  - Sozialmed. Zentrum Ost - Donauspital, Vienna
- Hungary (9):
  - SZTE AOK Borgyogyaszati es Allergologiai Klinika, Szeged, Csongrád megye
  - Debreceni Egyetem Klinikai Kozpont Borgyogyaszati Klinika, Debrecen, Hajdú-Bihar
  - Trial Pharma Kft., Püspökladány, Hajdú-Bihar
  - Allergo-Derm Bakos Kft, Szolnok, Jász-Nagykun-Szolnok
  - UNO Medical Trials Kft., Budapest
  - Kaposi Mor Oktato Korhaz, Kaposvár
  - Oroshaza Varosi Onkormanyzat Korhaza, Orosháza
  - Markusovszky Korhaz, Szombathely
  - MedMare Bt, Veszprém
- Israel (6):
  - Haemek Medical Center- Dermatology, Afula
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center - Ein Karem, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (16):
  - Yanagihara dermatology clinic, Ainokawa, Ichikawa-shi, Chiba
  - Kurume University Hospital, Kurume, Fukuoka
  - Sapporo Skin Clinic, Sapporo, Hokkaido
  - Tokyo Medical University Ibaraki Medical Center, Inashiki-gun, Ibaraki
  - Nomura Dermatology Clinic, Yokohama, Kanagawa
  - Noguchi Dermatology, Kashima-machi, Kamimashiki-gun, Kumamoto
  - Osaka Habikino Medical Center, Habikino, Osaka
  - Yoshioka Dermatology Clinic, Neyagawa, Osaka
  - Sanrui Dermatology Clinic, Ohmiya-ku,Saitama-shi, Saitama
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Tokyo Teishin Hospital, Chiyoda-Ku, Tokyo
  - Naoko Dermatology Clinic, Setagaya-ku, Tokyo
  - Yamate Dermatological Clinic, Shinjuku, Tokyo
  - Tachikawa Dermatology Clinic, Tachikawa-shi, Tokyo
  - Gifu University Hospital, Gifu
  - Osaka City University Hospital, Osaka
- Poland (10):
  - NZOZ Specjalistyczna Przychodnia Dermatologiczna Specderm, Bialystok
  - Centrum Badan Klinicznych, PI House, Gdansk
  - Centrum Medyczne Angelius Provita, Katowice
  - Barbara Rewerska DIAMOND CLINIC, Krakow
  - "Dermed" Centrum Medyczne Sp. z o.o., Lodz
  - Miejski Szpital Zespolony w Olsztynie, Olsztyn
  - DermoDent, Centrum Medyczne Czajkowscy, Osielsko
  - LASER CLINIC S.C. Dr Tomasz Kochanowski, Dr Andrzej Krolicki, Szczecin
  - Centralny Szpital Kliniczny MSW, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
- South Korea (7):
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Korea
  - Severance Hospital Yonsei University Health System, Seoul
  - Konkuk University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Chungang University Hospital, Seoul
  - Hallym University of Medicine, Seoul
- Spain (9):
  - Hospital Germans Trias i Pujol, Barcelona, Badalona
  - Hospital De Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Clinica Universitaria De Navarra, Pamplona, Navarre
  - Hospital General Universitario Alicante, Alicante
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Centro de Especialidades Mollabao, Pontevedra
- Switzerland (4):
  - CHUV Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - Inselspital Bern, Bern
  - HUG-Hôpitaux Universitaires de Genève, Geneva
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Katoh N, Takita Y, Isaka Y, Nishikawa A, Torisu-Itakura H, Saeki H. Pooled Safety Analysis of Baricitinib in Adult Participants with Atopic Dermatitis in the Japanese Subpopulation from Six Randomized Clinical Trials. Dermatol Ther (Heidelb). 2022 Dec;12(12):2765-2779. doi: 10.1007/s13555-022-00828-5. Epub 2022 Oct 18. PMID 36255569
- [Derived] Silverberg JI, DeLozier A, Sun L, Thyssen JP, Kim B, Yosipovitch G, Nunes FP, Gugiu PC, Doll HA, Eichenfield LF. Psychometric properties of the itch numeric rating scale, skin pain numeric rating scale, and atopic dermatitis sleep scale in adult patients with moderate-to-severe atopic dermatitis. Health Qual Life Outcomes. 2021 Oct 23;19(1):247. doi: 10.1186/s12955-021-01877-8. PMID 34688290
- [Derived] Thyssen JP, Buhl T, Fernandez-Penas P, Kabashima K, Chen S, Lu N, DeLozier AM, Casillas M, Stander S. Baricitinib Rapidly Improves Skin Pain Resulting in Improved Quality of Life for Patients with Atopic Dermatitis: Analyses from BREEZE-AD1, 2, and 7. Dermatol Ther (Heidelb). 2021 Oct;11(5):1599-1611. doi: 10.1007/s13555-021-00577-x. Epub 2021 Jul 18. PMID 34275122
- [Derived] Buhl T, Rosmarin D, Serra-Baldrich E, Fernandez-Penas P, Igarashi A, Konstantinou MP, Chen S, Lu N, Pierce E, Casillas M. Itch and Sleep Improvements with Baricitinib in Patients with Atopic Dermatitis: A Post Hoc Analysis of 3 Phase 3 Studies. Dermatol Ther (Heidelb). 2021 Jun;11(3):971-982. doi: 10.1007/s13555-021-00534-8. Epub 2021 Apr 25. PMID 33899152
- [Derived] King B, Maari C, Lain E, Silverberg JI, Issa M, Holzwarth K, Brinker D, Cardillo T, Nunes FP, Simpson EL. Extended Safety Analysis of Baricitinib 2 mg in Adult Patients with Atopic Dermatitis: An Integrated Analysis from Eight Randomized Clinical Trials. Am J Clin Dermatol. 2021 May;22(3):395-405. doi: 10.1007/s40257-021-00602-x. Epub 2021 Apr 7. PMID 33826132
- [Derived] Reich K, DeLozier AM, Nunes FP, Thyssen JP, Eichenfield LF, Wollenberg A, Ross Terres JA, Watts SD, Chen YF, Simpson EL, Silverberg JI. Baricitinib improves symptoms in patients with moderate-to-severe atopic dermatitis and inadequate response to topical corticosteroids: patient-reported outcomes from two randomized monotherapy phase III trials. J Dermatolog Treat. 2022 May;33(3):1521-1530. doi: 10.1080/09546634.2020.1839008. Epub 2020 Nov 22. PMID 33222559
- See also: A Study of Baricitinib (LY3009104) in Adults With Moderate to Severe Atopic Dermatitis (Eczema) (BREEZE-AD2) — https://www.lillytrialguide.com/en-US/studies/eczema/JAHM#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed double blind treatment phase had option to enter extension study I4V-MC-JAHN (NCT03334435).
Groups:
- 1mg Baricitinib: 1 milligram (mg) Baricitinib administered orally once daily.
- 2mg Baricitinib: 2mg Baricitinib administered orally once daily.
- 4mg Baricitinib: 4mg Baricitinib administered orally once daily.
Period: Overall Study
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Started | 244 | 125 | 123 | 123
Received at Least One Dose of Study Drug | 244 | 124 | 123 | 123
Completed | 225 | 115 | 113 | 117
Not Completed | 19 | 10 | 10 | 6
Not completed — Adverse Event | 1 | 3 | 2 | 2
Not completed — Lack of Efficacy | 10 | 2 | 7 | 3
Not completed — Withdrawal by Subject | 8 | 3 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Inability to obtain laboratory samples | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib | Total
Number analyzed (Participants) | 244 | 125 | 123 | 123 | 615
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 235 | 124 | 118 | 119 | 596
  >=65 years | 9 | 1 | 5 | 4 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 45 | 58 | 41 | 234
  Male | 154 | 80 | 65 | 82 | 381
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 72 | 36 | 37 | 38 | 183
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 169 | 85 | 85 | 82 | 421
  More than one race | 3 | 3 | 1 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 28 | 14 | 13 | 12 | 67
  South Korea | 24 | 11 | 11 | 9 | 55
  Austria | 13 | 7 | 4 | 7 | 31
  Hungary | 23 | 10 | 11 | 8 | 52
  Japan | 45 | 22 | 22 | 23 | 112
  Poland | 41 | 27 | 21 | 29 | 118
  Israel | 12 | 7 | 6 | 9 | 34
  Australia | 24 | 14 | 15 | 14 | 67
  Switzerland | 13 | 5 | 5 | 2 | 25
  Spain | 21 | 8 | 15 | 10 | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) of 0 or 1 With a ≥ 2 Point Improvement (Placebo, 2mg and 4mg Baricitinib)
Description: The IGA measures the investigator's global assessment of the participants overall severity of their atopic dermatitis (AD), based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: 16 Weeks
Population: All participants randomized to placebo, 2mg, or 4mg of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 244 | 123 | 123
percentage of participants | 4.5 | 10.6 | 13.8
Statistical Analysis 1: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p = 0.026, Regression, Logistic; Odds Ratio (OR) = 2.58, 95% CI 2-sided [1.12 to 5.92]
Statistical Analysis 2: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 3.64, 95% CI 2-sided [1.64 to 8.05]

2. Secondary Outcome: Percentage of Participants Achieving IGA of 0 or 1 With a ≥ 2 Point Improvement (Placebo, 1mg Baricitinib)
Description: The IGA measures the investigator's global assessment of the participants overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: 16 Weeks
Population: All participants randomized to placebo or 1mg of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1mg Baricitinib
Number analyzed (Participants) | 244 | 125
percentage of participants | 4.5 | 8.8
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.085, Regression, Logistic; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.90 to 5.02]

3. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index 75 (EASI75)
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2 and 3. The final EASI score is obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI75 is defined as a ≥ 75% improvement from baseline in the EASI score.
Time Frame: 16 Weeks
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Groups:
- 1mg Baricitinib: 1mg Baricitinib administered orally once daily.
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 244 | 125 | 123 | 123
percentage of participants | 6.1 | 12.8 | 17.9 | 21.1
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.024, Regression, Logistic; Odds Ratio (OR) = 2.35, 95% CI 2-sided [1.12 to 4.93]
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.49, 95% CI 2-sided [1.73 to 7.04]
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.41, 95% CI 2-sided [2.22 to 8.76]

4. Secondary Outcome: Percentage of Participants Achieving EASI90
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100%) and the severity of 4 clinical signs (1) erythema, (2)edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2 and 3. The final EASI score is obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI90 is defined as a ≥ 90% improvement from baseline in the EASI score.
Time Frame: 16 Weeks
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 244 | 125 | 123 | 123
percentage of participants | 2.5 | 6.4 | 8.9 | 13.0
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.053, Regression, Logistic; Odds Ratio (OR) = 2.80, 95% CI 2-sided [0.99 to 7.97]
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p = 0.007, Regression, Logistic; Odds Ratio (OR) = 3.87, 95% CI 2-sided [1.44 to 10.41]
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.20, 95% CI 2-sided [2.42 to 15.91]

5. Secondary Outcome: Percent Change From Baseline on EASI Score
Description: The EASI assesses objective physician estimates of 2 dimensions of AD - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs (1) erythema (2)edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2 and 3. The final EASI score is obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  Least Square (LS) Means were calculated using a mixed model repeated measures (MMRM) model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants who had a week 16 EASI data.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 52 | 34 | 40 | 49
Percent Change | -28.91 (4.32) | -41.68 (5.33) | -54.80 (4.99) | -54.88 (4.56)
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.062, Mixed Models Analysis; Mean Difference (Net) = -12.76, 95% CI 2-sided [-26.19 to 0.66], Standard Error of Mean 6.81
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -25.89, 95% CI 2-sided [-38.78 to -12.99], Standard Error of Mean 6.54
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -25.97, 95% CI 2-sided [-38.29 to -13.65], Standard Error of Mean 6.24

6. Secondary Outcome: Percentage of Participants Achieving SCORing Atopic Dermatitis 75 (SCORAD75)
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable Itching or lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease. The SCORAD75 responder is defined as a participant who achieves a ≥ 75% improvement from baseline in the SCORAD score.
Time Frame: 16 Weeks
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 244 | 125 | 123 | 123
percentage of participants | 1.6 | 4.8 | 7.3 | 11.4
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.086, Regression, Logistic; Odds Ratio (OR) = 2.90, 95% CI 2-sided [0.86 to 9.76]
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 4.95, 95% CI 2-sided [1.58 to 15.49]
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.40, 95% CI 2-sided [2.51 to 21.83]

7. Secondary Outcome: Percentage of Participants Achieving a 4-Point Improvement in Itch Numeric Rating Scale (NRS)
Description: The Itch Numeric Rating Scale (NRS) is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participants itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours.
Time Frame: 16 Weeks
Population: All randomized participants with a baseline Itch NRS score ≥ 4.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 213 | 100 | 106 | 107
percentage of participants | 4.7 | 6.0 | 15.1 | 18.7
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.505, Regression, Logistic; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.51 to 3.87]
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 3.64, 95% CI 2-sided [1.60 to 8.27]
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.91, 95% CI 2-sided [2.22 to 10.86]

8. Secondary Outcome: Change From Baseline in the Score of Item 2 of the Atopic Dermatitis Sleep Scale (ADSS)
Description: Atopic Dermatitis Sleep Scale (ADSS) is a 3-item, participant-administered questionnaire developed to assess the impact of itch on sleep including difficulty falling asleep, frequency of waking, and difficulty getting back to sleep last night. Item 2, frequency of waking last night is reported by selecting the number of times they woke up each night, ranging from 0 to 29 times, where the higher a number indicates a worse outcome. The ADSS is designed to be completed daily, using a daily diary, with respondents thinking about sleep "last night." Each item is scored individually.
  LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by- visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with a Week 16 ADSS Item 2 (frequency of waking) data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 208 | 103 | 105 | 112
units on a scale | -0.8 (0.09) | -1.10 (0.12) | -1.21 (0.12) | -1.38 (0.12)
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.074, Mixed Models Analysis; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.57 to 0.03], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p = 0.011, Mixed Models Analysis; Mean Difference (Net) = -0.38, 95% CI 2-sided [-0.68 to -0.09], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.55, 95% CI 2-sided [-0.84 to -0.26], Standard Error of Mean 0.15

9. Secondary Outcome: Change From Baseline in Skin Pain NRS
Description: Skin Pain NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no pain" and 10 representing "worst pain imaginable." Overall severity of a participant's skin pain is indicated by selecting the number, using a daily diary, that best describes the worst level of skin pain in the past 24 hours.
  LSMean was calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with a Week 16 Skin Pain NRS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 49 | 31 | 38 | 47
units on a scale | -0.86 (0.26) | -1.09 (0.32) | -2.61 (0.30) | -2.49 (0.28)
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.580, Mixed Models Analysis; Mean Difference (Net) = -0.23, 95% CI 2-sided [-1.05 to 0.59], Standard Error of Mean 0.41
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.75, 95% CI 2-sided [-2.54 to -0.96], Standard Error of Mean 0.40
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.62, 95% CI 2-sided [-2.37 to -0.87], Standard Error of Mean 0.38

10. Secondary Outcome: Percentage of Participants Achieving EASI50
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs (1) erythema, (2)edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2 and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI 50 is defined as ≥50% improvement from baseline in EASI score.
Time Frame: 16 Weeks
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Groups:
- 2mg Bariciitnib: 2mg Baricitinib administered orally once daily.
Arm/Group | Placebo | 1mg Baricitinib | 2mg Bariciitnib | 4mg Baricitinib
Number analyzed (Participants) | 244 | 125 | 123 | 123
percentage of participants | 12.3 | 18.4 | 27.6 | 29.3
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.094, Regression, Logistic; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.92 to 3.04]
Statistical Analysis 2: Comparison: Placebo vs 2mg Bariciitnib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.91, 95% CI 2-sided [1.65 to 5.11]
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.15, 95% CI 2-sided [1.80 to 5.51]

11. Secondary Outcome: Percentage of Participants Achieving IGA of 0
Description: as for outcome 2
Time Frame: 16 Weeks
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 244 | 125 | 123 | 123
percentage of participants | 1.6 | 2.4 | 4.1 | 4.1
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.528, Regression, Logistic; Odds Ratio (OR) = 1.57, 95% CI 2-sided [0.39 to 6.31]
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p = 0.142, Regression, Logistic; Odds Ratio (OR) = 2.56, 95% CI 2-sided [0.73 to 8.95]
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p = 0.123, Regression, Logistic; Odds Ratio (OR) = 2.68, 95% CI 2-sided [0.77 to 9.37]

12. Secondary Outcome: Change From Baseline in SCORAD
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable itching or lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease. LSMeans was calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, & treatment-by-visit-interaction as fixed categorical effects. Baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with a Week 16 SCORAD data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 52 | 34 | 40 | 49
units on a scale | -13.35 (2.31) | -20.23 (2.84) | -27.83 (2.62) | -27.50 (2.41)
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.059, Mixed Models Analysis; LSMean Difference = -6.88, 95% CI 2-sided [-14.03 to 0.28], Standard Error of Mean 3.63
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -14.48, 95% CI 2-sided [-21.32 to -7.63], Standard Error of Mean 3.47
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -14.15, 95% CI 2-sided [-20.69 to -7.61], Standard Error of Mean 3.32

13. Secondary Outcome: Percentage of Participants Achieving SCORAD90
Description: The SCORAD index uses the rule of nines to assess disease extent and evaluates 6 clinical characteristics to determine disease severity: (1) erythema, (2) edema/papulation, (3) oozing/crusts, (4) excoriation, (5) lichenification, and (6) dryness on a scale of 0 to 3 (0=absence, 1=mild, 2=moderate, 3=severe). The SCORAD index also assesses subjective symptoms of pruritus and sleep loss with VAS where 0 is no itching or no trouble sleeping and 10 is unbearable itching or lot of trouble sleeping. These 3 aspects: extent of disease (A: 0-1-2), disease severity (B: 0-18), & subjective symptoms (C: 0-20) combine using A/5 + 7*B/2+ C to give a maximum possible score of 103, where 0 = no disease and 103 = severe disease.
  SCORAD90 defined as a ≥ 90% improvement from baseline in the SCORAD score.
Time Frame: 16 Weeks
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 244 | 125 | 123 | 123
percentage of participants | 1.2 | 3.2 | 4.1 | 4.9
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.193, Regression, Logistic; Odds Ratio (OR) = 2.55, 95% CI 2-sided [0.62 to 10.45]
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p = 0.042, Mixed Models Analysis; Odds Ratio (OR) = 4.10, 95% CI 2-sided [1.05 to 16.03]
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p = 0.044, Regression, Logistic; Odds Ratio (OR) = 3.89, 95% CI 2-sided [1.04 to 14.57]

14. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) Affected
Description: Body surface area affected by AD will be assessed for 4 separate body regions and is collected as part of the EASI assessment: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). Each body region will be assessed for disease extent ranging from 0% to 100% involvement. The overall total percentage will be reported based off of all 4 body regions combined, after applying specific multipliers to the different body regions to account for the percent of the total BSA represented by each of the 4 regions.
  Use the percentage of skin affected for each region (0 to 100%) in EASI as follows:
  BSA Total = 0.1*BSAhead and neck + 0.3*BSAtrunk + 0.2* BSAupper limbs + 0.4*BSAlower limbs.
  LSMean were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 BSA data.
Measure: Median (Standard Error); unit: unit on a scale
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 52 | 34 | 40 | 49
unit on a scale | 12.82 (2.07) | -18.98 (2.53) | -22.12 (2.37) | -23.98 (2.17)
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.058, Mixed Models Analysis; LSMean Difference = -6.16, 95% CI 2-sided [-12.53 to 0.21], Standard Error of Mean 3.23
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p = 0.003, Mixed Models Analysis; LSMean Difference = -9.30, 95% CI 2-sided [-15.42 to -3.18], Standard Error of Mean 3.10
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -11.16, 95% CI 2-sided [-17.03 to -5.30], Standard Error of Mean 2.98

15. Secondary Outcome: Percentage of Participants Developing Skin Infections Requiring Antibiotic Treatment
Description: Percentage of participants developing skin infections requiring antibiotic treatment.
Time Frame: 16 Weeks
Population: All randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 244 | 124 | 123 | 123
Percentage of participants | 7.8 | 4.8 | 7.3 | 4.9
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.189, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p = 1, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p = 0.383, Fisher Exact

16. Secondary Outcome: Percent Change From Baseline in Itch NRS
Description: The Itch NRS is a participant-administered, 11-point horizontal scale, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching is indicated by selecting the number, using a daily diary, that best describes the worst level of itching in the past 24 hours.
  LSMean were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, & treatment-by-visit-interaction as fixed categorical effects. Baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with week 16 Itch NRS data.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 48 | 31 | 38 | 47
Percent Change | -16.58 (5.45) | -31.39 (6.61) | 47.24 (6.10) | 46.87 (5.43)
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.081, Mixed Models Analysis; LSMean Difference = -14.80, 95% CI 2-sided [-31.45 to 1.85], Standard Error of Mean 8.46
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -30.66, 95% CI 2-sided [-46.62 to -14.70], Standard Error of Mean 8.11
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -30.28, 95% CI 2-sided [-45.29 to -15.27], Standard Error of Mean 7.63

17. Secondary Outcome: Change From Baseline in the Total Score of the Patient Oriented Eczema Measure (POEM)
Description: The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) on a scale ranging from 0-4 (0 = no days, 1 = 1-2 days, 2 = 3-4 days, 3 = 5-6 days, 4 = everyday). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). High scores are indicative of more severe disease and poor quality of life.
  LSMean were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, & treatment-by-visit-interaction as fixed categorical effects. Baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with week 16 POEM data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 52 | 34 | 40 | 48
units on a scale | -1.48 (0.84) | -3.85 (1.04) | -7.06 (0.96) | -7.56 (0.88)
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.075, Mixed Models Analysis; LSMean Difference = -2.36, 95% CI 2-sided [-4.97 to 0.24], Standard Error of Mean 1.32
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -5.58, 95% CI 2-sided [-8.07 to -3.08], Standard Error of Mean 1.27
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -6.07, 95% CI 2-sided [-8.47 to -3.68], Standard Error of Mean 1.21

18. Secondary Outcome: Change From Baseline in the Patient Global Impression of Severity-Atopic Dermatitis (PGI-S-AD) Score
Description: The PGI-S-AD asked the participant to evaluate the severity of the disease at that point in time on a single-item, 5-point scale, using a daily diary. The same category labels used in the Physician's Global Assessment were used for the PGI-S-AD, ie, "(0) no symptoms", "(1) very mild", "(2) mild" "(3) moderate", and "(4) severe." LS Means were calculated using a MMRM model with treatment, region, baseline disease severity (IGA), visit, and treatment-by-visit-interaction as fixed categorical effects and baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 PGI-S-AD data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 49 | 31 | 38 | 47
units on a scale | -0.27 (0.11) | -0.53 (0.14) | -0.88 (0.13) | -0.96 (0.12)
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.130, Mixed Models Analysis; LSMean Difference = -0.27, 95% CI 2-sided [-0.61 to 0.08], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -0.61, 95% CI 2-sided [-0.94 to -0.28], Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -0.69, 95% CI 2-sided [-1.00 to -0.38], Standard Error of Mean 0.16

19. Secondary Outcome: Change From Baseline on the Hospital Anxiety and Depression Scale (HADS)
Description: The HADS is a participant-rated instrument used to assess both anxiety and depression. This instrument consists of 14 items questionnaire, each item is rated on a 4-point scale, giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7, 'normal.
  LSMean were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, & treatment-by-visit-interaction as fixed categorical effects. Baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with Week 16 HADS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 52 | 34 | 40 | 48
units on a scale
  Anxiety | -0.99 (0.33) | -1.93 (0.40) | -1.92 (0.38) | -2.30 (0.35)
  Depression | -0.28 (0.32) | -0.78 (0.40) | -0.99 (0.37) | -1.46 (0.35)
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; HADS Anxiety; Test type: Superiority; p = 0.067, Mixed Models Analysis; LSMean Difference = -0.94, 95% CI 2-sided [-1.95 to 0.07], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; HADS Anxiety; Test type: Superiority; p = 0.060, Mixed Models Analysis; LSMean Difference = -0.93, 95% CI 2-sided [-1.89 to 0.04], Standard Error of Mean 0.49
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; HADS Anxiety; Test type: Superiority; p = 0.006, Mixed Models Analysis; LSMean Difference = -1.30, 95% CI 2-sided [-2.23 to -0.38], Standard Error of Mean 0.47
Statistical Analysis 4: Comparison: Placebo vs 1mg Baricitinib; HADS Depression; Test type: Superiority; p = 0.321, Mixed Models Analysis; LSMean Difference = -0.50, 95% CI 2-sided [-1.50 to 0.49], Standard Error of Mean 0.51
Statistical Analysis 5: Comparison: Placebo vs 2mg Baricitinib; HADS Depression; Test type: Superiority; p = 0.143, Mixed Models Analysis; LSMean Difference = -0.71, 95% CI 2-sided [-1.67 to 0.24], Standard Error of Mean 0.49
Statistical Analysis 6: Comparison: Placebo vs 4mg Baricitinib; HADS Depression; Test type: Superiority; p = 0.012, Mixed Models Analysis; LSMean Difference = -1.18, 95% CI 2-sided [-2.11 to -0.26], Standard Error of Mean 0.47

20. Secondary Outcome: Change From Baseline on the Dermatology Life Quality Index (DLQI)
Description: The DLQI is a simple, participant-administered, 10 question, validated, quality-of-life questionnaire that covers 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The recall period of this scale is over the last "week." Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as "0." Scores range from 0 to 30 (less to more impairment), and a 4-point change from baseline is considered as the minimal clinically important difference threshold.
  LSMean were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, & treatment-by-visit-interaction as fixed categorical effects. Baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with week 16 DLQI data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Participants received placebo orally once daily for 16 weeks.
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 52 | 34 | 40 | 48
units on a scale | -3.35 (0.62) | -5.11 (0.76) | -7.44 (0.71) | -7.56 (0.66)
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.071, Mixed Models Analysis; LSMean Difference = -1.76, 95% CI 2-sided [-3.67 to 0.15], Standard Error of Mean 0.97
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -4.09, 95% CI 2-sided [-5.92 to -2.26], Standard Error of Mean 0.93
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -4.22, 95% CI 2-sided [-5.98 to -2.45], Standard Error of Mean 0.90

21. Secondary Outcome: Change From Baseline on the Work Productivity and Activity Impairment - Atopic Dermatitis (WPAI-AD) Questionnaire
Description: The WPAI-AD participant questionnaire was developed to measure the effect of general health and symptom severity on work productivity and regular activities in the 7 days prior to the visit. The WPAI-AD consists of 6 items grouped in 4 domains: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment, that range from 0% to 100%, with higher values indicating greater impairment. LSMean were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, & treatment-by-visit-interaction as fixed categorical effects. Baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with week 16 WPAI-AD data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 52 | 34 | 39 | 49
units on a scale
  Absenteeism: number analyzed (Participants) | 25 | 21 | 22 | 33
  Absenteeism | -4.40 (3.45) | -5.31 (3.91) | -3.39 (3.68) | 0.76 (3.08)
  Presentisms: number analyzed (Participants) | 23 | 21 | 22 | 32
  Presentisms | -6.15 (3.87) | -9.27 (4.08) | -19.71 (3.90) | -19.28 (3.37)
  Work Productivity Loss: number analyzed (Participants) | 23 | 21 | 22 | 32
  Work Productivity Loss | -7.15 (4.65) | -8.96 (4.86) | -16.63 (4.65) | -16.28 (3.96)
  Activities Impairment | -8.94 (2.74) | -11.21 (3.34) | -23.25 (3.12) | -23.41 (2.82)
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Percentage of Absenteeism Change from Baseline; Test type: Superiority; p = 0.861, Mixed Models Analysis; LSMean Difference = -0.91, 95% CI 2-sided [-11.16 to 9.34], Standard Error of Mean 5.17
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Percentage of Absenteeism Change from Baseline; Test type: Superiority; p = 0.841, Mixed Models Analysis — Absenteeism; LSMean Difference = 1.01, 95% CI 2-sided [-8.94 to 10.97], Standard Error of Mean 5.03
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Percentage of Absenteeism Change from Baseline; Test type: Superiority; p = 0.264, Mixed Models Analysis; LSMean Difference = 5.16, 95% CI 2-sided [-3.95 to 14.26], Standard Error of Mean 4.60
Statistical Analysis 4: Comparison: Placebo vs 1mg Baricitinib; Percentage of Presenteeism (Reduced Productivity While at Work) Change from Baseline; Test type: Superiority; p = 0.580, Mixed Models Analysis; LSMean Difference = -3.12, 95% CI 2-sided [-14.26 to 8.02], Standard Error of Mean 5.63
Statistical Analysis 5: Comparison: Placebo vs 2mg Baricitinib; Percentage of Presenteeism (Reduced Productivity While at Work) Change from Baseline; Test type: Superiority; p = 0.015, Mixed Models Analysis; LSMean Difference = -13.56, 95% CI 2-sided [-24.45 to -2.86], Standard Error of Mean 5.50
Statistical Analysis 6: Comparison: Placebo vs 4mg Baricitinib; Percentage of Presenteeism (Reduced Productivity While at Work) Change from Baseline; Test type: Superiority; p = 0.011, Mixed Models Analysis; LSMean Difference = -13.13, 95% CI 2-sided [-23.20 to -3.06], Standard Error of Mean 5.08
Statistical Analysis 7: Comparison: Placebo vs 1mg Baricitinib; Work Productivity Loss (Percentage Overall Work Impairment/Absenteeism Plus Presenteeism) Change from Baseline; Test type: Superiority; p = 0.788, Mixed Models Analysis; LSMean Difference = -1.81, 95% CI 2-sided [-15.12 to 11.49], Standard Error of Mean 6.71
Statistical Analysis 8: Comparison: Placebo vs 2mg Baricitinib; Work Productivity Loss (Percentage Overall Work Impairment/Absenteeism Plus Presenteeism) Change from Baseline; Test type: Superiority; p = 0.152, Mixed Models Analysis; LSMean Difference = -9.48, 95% CI 2-sided [-22.51 to 3.55], Standard Error of Mean 6.57
Statistical Analysis 9: Comparison: Placebo vs 4mg Baricitinib; Work Productivity Loss (Percentage Overall Work Impairment/Absenteeism Plus Presenteeism) Change from Baseline; Test type: Superiority — Overall Work Impairment; p = 0.135, Mixed Models Analysis; LSMean Difference = -9.13, 95% CI 2-sided [-21.17 to 2.90], Standard Error of Mean 6.07
Statistical Analysis 10: Comparison: Placebo vs 1mg Baricitinib; Percentage of Activity Impairment Change from Baseline; Test type: Superiority; p = 0.595, Mixed Models Analysis; LSMean Difference = -2.26, 95% CI 2-sided [-10.65 to 6.12], Standard Error of Mean 4.25
Statistical Analysis 11: Comparison: Placebo vs 2mg Baricitinib; Percentage of Activity Impairment Change from Baseline; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -14.30, 95% CI 2-sided [-22.43 to -6.17], Standard Error of Mean 4.12
Statistical Analysis 12: Comparison: Placebo vs 4mg Baricitinib; Percentage of Activity Impairment Change from Baseline; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -14.47, 95% CI 2-sided [-22.11 to -6.83], Standard Error of Mean 3.88

22. Secondary Outcome: Change From Baseline on the European Quality of Life-5 Dimensions 5 Levels (EQ-5D-5L) Index Score United States and United Kingdom Algorithm
Description: EQ-5D-5L is a 2-part measurement. The first part is comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.594 to 1, and the United States (US) algorithm, with scores ranging from -0.109 to 1. A higher score indicates better health state.
  LSMean were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, & treatment-by-visit-interaction as fixed categorical effects. Baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with week 16 EQ-5D-5L health state index US & UK data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 52 | 34 | 39 | 49
units on a scale
  Health State Index Score (US Algorithm) | 0.02 (0.02) | 0.05 (0.02) | 0.10 (0.02) | 0.10 (0.02)
  Health State Index Score (UK Algorithm) | 0.03 (0.02) | 0.06 (0.03) | 0.14 (0.02) | 0.14 (0.02)
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Health State Index Score (US Algorithm); Test type: Superiority; p = 0.295, Mixed Models Analysis; LSMean Difference = 0.02, 95% CI 2-sided [-0.02 to 0.07], Standard Error of Mean 0.02
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Health State Index Score (US Algorithm); Test type: Superiority; p = 0.001, Mixed Models Analysis; LSMean Difference = 0.08, 95% CI 2-sided [0.03 to 0.12], Standard Error of Mean 0.02
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Health State Index Score (US Algorithm); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = 0.08, 95% CI 2-sided [0.03 to 0.12], Standard Error of Mean 0.02
Statistical Analysis 4: Comparison: Placebo vs 1mg Baricitinib; Health State Index Score (UK Algorithm); Test type: Superiority; p = 0.334, Mixed Models Analysis; LSMean Difference = 0.03, 95% CI 2-sided [-0.03 to 0.10], Standard Error of Mean 0.03
Statistical Analysis 5: Comparison: Placebo vs 2mg Baricitinib; Health State Index Score (UK Algorithm); Test type: Superiority; p = 0.001, Mixed Models Analysis; LSMean Difference = 0.11, 95% CI 2-sided [0.04 to 0.17], Standard Error of Mean 0.03
Statistical Analysis 6: Comparison: Placebo vs 4mg Baricitinib; Health State Index Score (UK Algorithm); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = 0.11, 95% CI 2-sided [0.05 to 0.17], Standard Error of Mean 0.03

23. Secondary Outcome: Change From Baseline on the European Quality of Life-5 Dimensions 5 Levels (EQ-5D-5L) Visual Analog Score (VAS)
Description: EQ-5D-5L is a 2-part measurement. The second part is assessed using a visual analog scale (VAS) that ranged from 0 to 100 millimeter (mm), where 0 is the worst health you can imagine and 100 is the best health you can imagine.
  LSMean were calculated using MMRM model with treatment, region, baseline disease severity (IGA), visit, & treatment-by-visit-interaction as fixed categorical effects. Baseline and baseline-by-visit-interaction as fixed continuous effects.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants with week 16 EQ-5D-5L VAS data.
Measure: Least Squares Mean (Standard Error); unit: Millimeter (mm)
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 52 | 34 | 39 | 49
Millimeter (mm) | 2.34 (2.22) | 2.75 (2.71) | 10.54 (2.53) | 11.16 (2.30)
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; EQ-5D-5L VAS Score; Test type: Superiority; p = 0.907, Mixed Models Analysis; LSMean Difference = 0.40, 95% CI 2-sided [-6.44 to 7.25], Standard Error of Mean 3.47
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; EQ-5D-5L VAS Score; Test type: Superiority; p = 0.015, Mixed Models Analysis; LSMean Difference = 8.19, 95% CI 2-sided [1.63 to 14.76], Standard Error of Mean 3.33
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; EQ-5D-5L VAS Score; Test type: Superiority; p = 0.006, Mixed Models Analysis; LSMean Difference = 8.82, 95% CI 2-sided [2.62 to 15.01], Standard Error of Mean 3.14

24. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) of 0 or 1 With a ≥ 2 Point Improvement
Description: as for outcome 2
Time Frame: 4 Weeks
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
Number analyzed (Participants) | 244 | 125 | 123 | 123
percentage of participants | 3.7 | 3.2 | 8.1 | 15.4
Statistical Analysis 1: Comparison: Placebo vs 1mg Baricitinib; Test type: Superiority; p = 0.905, Regression, Logistic; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.30 to 2.93]
Statistical Analysis 2: Comparison: Placebo vs 2mg Baricitinib; Test type: Superiority; p = 0.064, Regression, Logistic; Odds Ratio (OR) = 2.37, 95% CI 2-sided [0.95 to 5.92]
Statistical Analysis 3: Comparison: Placebo vs 4mg Baricitinib; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.14, 95% CI 2-sided [2.25 to 11.74]

ADVERSE EVENTS:
Time Frame: Baseline to end of study (Up to 20 weeks)
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Placebo | 1mg Baricitinib | 2mg Baricitinib | 4mg Baricitinib
All-Cause Mortality (participants affected / at risk) | 0/244 | 0/124 | 0/123 | 0/123
Serious Adverse Events (participants affected / at risk) | 9/244 | 9/124 | 3/123 | 1/123
Other Adverse Events (participants affected / at risk) | 34/244 | 23/124 | 27/123 | 29/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=244) | 1mg Baricitinib (N=124) | 2mg Baricitinib (N=123) | 4mg Baricitinib (N=123)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema herpeticum (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Encephalitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=244) | 1mg Baricitinib (N=124) | 2mg Baricitinib (N=123) | 4mg Baricitinib (N=123)
Herpes simplex (Infections and infestations) | 2 (3) | 2 (2) | 7 (7) | 3 (3)
Nasopharyngitis (Infections and infestations) | 30 (33) | 13 (13) | 16 (16) | 10 (12)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 4 (4) | 1 (1) | 7 (7)
Headache (Nervous system disorders) | 5 (8) | 6 (6) | 9 (9) | 11 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT03334422/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT03334422/SAP_001.pdf